CLINICAL TRIAL: NCT03456713
Title: A Safety, Tolerability, and Pharmacokinetic Study of 1- and 2-mL Injections of LY3074828 Solution Using Investigational Pre-filled Syringes and Investigational Autoinjectors in Healthy Subjects
Brief Title: A Study of LY3074828 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16617; I6T-MC-AMAQ (Other: Eli Lilly and Company.)
Record Dates: First submitted 2018-03-05; First posted 2018-03-07 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: 250 mg LY3074828 (Reference) (Experimental): 250 mg LY3074828 administered subcutaneous (SC) as solution formulation in two prefilled syringes targeting a 5- to 10-second injection time for each injection on day 1.
  Interventions: Biological: LY3074828
- Part A: 250 mg LY3074828 (Test 1) (Experimental): 250 mg LY3074828 administered SC as solution formulation in a prefilled syringe targeting a 5- to 15-second injection time on day 1.
  Interventions: Biological: LY3074828
- Part B: 250 mg LY3074828 (Test 2 and Test 3) (Experimental): Test 2: 250 mg LY3074828 administered subcutaneous (SC) as solution formulation in an auto-injector at slow speed targeting an approximately 13-second injection time on day 1.
  Test 3: 250 mg LY3074828 administered subcutaneous (SC) as solution formulation in an auto-injector at fast speed targeting an approximately 5-second injection time on day 2.
  Interventions: Biological: LY3074828
- Part B: 125 mg LY3074828 (Test 4 and Test 5) (Experimental): Test 4: 125 mg LY3074828 administered SC as solution formulation in an auto-injector at slow speed targeting an approximately 7-second injection time on day 1.
  Test 5: 125 mg LY3074828 administered SC as solution formulation in an auto-injector at fast speed targeting an approximately 4.5-second injection time on day 2.
  Interventions: Biological: LY3074828

INTERVENTIONS:
Biological: LY3074828 — Administered SC

SUMMARY:
The purpose of this study is to look at the amount of the study drug, LY3074828, that gets into the blood stream and how long it takes the body to get rid of LY3074828, when given as a solution formulation in different devices. The tolerability of LY3074828 will also be evaluated and information about any side effects experienced will be collected.

Screening is required within 28 days prior to the start of the study. For each participant, the total duration of the clinical trial will be approximately 13 weeks, not including screening.

ELIGIBILITY:
Inclusion Criteria:

- Must be healthy male or female

Exclusion Criteria:

* Must not have an average weekly alcohol intake that exceeds 21 units/week (males) and 14 units/week (females)
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 1 month of screening, or intend to during the study
* Must not have been treated with steroids within 1 month of screening, or intend to during the study
* Must not be immunocompromised
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to Day 1
* Must not have significant allergies to humanised monoclonal antibodies
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or sever post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had a screening period of 28 days and residential period with a parallel 2 day Part A and a crossover 3 day Part B.
Period: Overall Study
Arm/Group | Part A: 250 mg LY3074828 (Reference) | Part A: 250 mg LY3074828 (Test 1) | Part B: 250 mg LY3074828 (Test 2 and Test 3) | Part B: 125 mg LY3074828 (Test 4 and Test 5)
Started | 18 | 18 | 18 | 18
Received at Least One Dose of Study Drug | 18 | 18 | 18 | 18
Completed | 17 | 18 | 18 | 18
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part B: 250 mg LY3074828 (Test 2 and Test 3): Test 2: 250 mg LY3074828 administered subcutaneous (SC) as solution formulation in an auto-injector at slow speed targeting an approximately 13-second injection time on day 1
  Test 3: 250 mg LY3074828 administered subcutaneous (SC) as solution formulation in an auto-injector at fast speed targeting an approximately 5-second injection time on day 2
- Part B: 125 mg LY3074828 (Test 4 and Test 5): Test 4: 125 mg LY3074828 administered SC as solution formulation in an auto-injector at slow speed targeting an approximately 7-second injection time on day 1
  Test 5: 125 mg LY3074828 administered SC as solution formulation in an auto-injector at fast speed targeting an approximately 4.5-second injection time on day 2.
- Total: Total of all reporting groups
Arm/Group | Part A: 250 mg LY3074828 (Reference) | Part A: 250 mg LY3074828 (Test 1) | Part B: 250 mg LY3074828 (Test 2 and Test 3) | Part B: 125 mg LY3074828 (Test 4 and Test 5) | Total
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 72
Age, Continuous [Mean (Standard Deviation); unit: years]
  Part A | 37.3 (12.7) | 33.9 (11.0) | NA (NA) — Row represents part A data. | NA (NA) — Row represents part A data. | 35.6 (11.8)
  Part B | NA (NA) — Row represents part B data. | NA (NA) — Row represents part B data. | 42.1 (12.3) | 47.2 (12.3) | 44.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 8 | 6 | 33
  Male | 9 | 8 | 10 | 12 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 3 | 6 | 17
  Not Hispanic or Latino | 12 | 16 | 15 | 12 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 6 | 5 | 26
  White | 10 | 10 | 10 | 10 | 40
  More than one race | 0 | 1 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 18 | 18 | 72

OUTCOME MEASURES:

1. Primary Outcome: Part A: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3074828
Description: Part A: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3074828
Time Frame: Day 1: 0, 2, 6; Day 2: 24; Day 4: 72; Day 8: 168; Day 11: 240; Day 15: 336; Day 22: 504; Day 29: 672; Day 43: 1008; Day 57: 1344; Day 71: 1680; Day 85: 2016 hours
Population: Part A: All randomized participants who received at least one dose of LY3074828 and have evaluable PK data. Per protocol only Part A data were analyzed for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliters (μg/mL)
Arm/Group | Part A: 250 mg LY3074828 (Reference) | Part A: 250 mg LY3074828 (Test 1)
Number analyzed (Participants) | 18 | 18
microgram per milliliters (μg/mL) | 14.4 (67) | 21.1 (34)
Statistical Analysis 1: Comparison: Part A: 250 mg LY3074828 (Reference) vs Part A: 250 mg LY3074828 (Test 1); Test type: Other; Ratio of geometric least squares mean = 1.47, 90% CI 2-sided [1.12 to 1.94]

2. Primary Outcome: Part A PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of LY3074828
Description: Part A PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of LY3074828
Time Frame: as for outcome 1
Population: All randomized participants who received at least one dose of LY3074828 and have evaluable PK data in Part A. Per protocol only Part A data were analyzed for PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*Day per Milliliters(μg*day/mL)
Arm/Group | Part A: 250 mg LY3074828 (Reference) | Part A: 250 mg LY3074828 (Test 1)
Number analyzed (Participants) | 14 | 18
Microgram*Day per Milliliters(μg*day/mL) | 240 (46) | 346 (33)
Statistical Analysis 1: Comparison: Part A: 250 mg LY3074828 (Reference) vs Part A: 250 mg LY3074828 (Test 1); Test type: Other; Ratio of geometric least squares mean = 1.44, 90% CI 2-sided [1.15 to 1.81]

3. Primary Outcome: Part A PK: Area Under the Concentration Versus Time Curve From Time Zero to Tlast (AUC[0-tlast]) of LY3074828
Description: Part A PK: Area Under the Concentration Versus Time Curve From Time Zero to tlast (AUC[0-tlast]) of LY3074828
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*Day per Milliliters(μg*day/mL)
Arm/Group | Part A: 250 mg LY3074828 (Reference) | Part A: 250 mg LY3074828 (Test 1)
Number analyzed (Participants) | 17 | 18
Microgram*Day per Milliliters(μg*day/mL) | 205 (54) | 341 (33)
Statistical Analysis 1: Comparison: Part A: 250 mg LY3074828 (Reference) vs Part A: 250 mg LY3074828 (Test 1); Test type: Other; Ratio of geometric least squares mean = 1.66, 90% CI 2-sided [1.31 to 2.11]

4. Primary Outcome: Part A: Short Form McGill Pain Questionnaire (SF-MPQ) Total Score (Including Visual Analog Scale (VAS ) Score)
Description: Pain was assessed by the SF-MPQ and quantified using the validated VAS where 0mm represented "no pain" and 100mm represented "worst possible pain". The SF-MPQ total score ranges from 0 to 45 (the higher the total score, the more pain experienced). Least Squares (LS) mean was calculated using linear fixed-effects model with treatment (Reference or Test 1) as a fixed effect. Model: Log (Score+1) = Treatment + Random Error.
Time Frame: Day 1, 0 hour
Population: All participants who received a dose of LY3074828 whether or not they completed all protocol requirements.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: units on a scale
Groups:
- Part A: 250 mg LY3074828 (Reference): 250 mg LY3074828 administered subcutaneous (SC) as solution, formulation in two prefilled syringes on day 1.
- Part A: 250 mg LY3074828 (Test 1): 250 mg LY3074828 solution formulation in a prefilled syringe, administered as a SC injection on day 1.
Arm/Group | Part A: 250 mg LY3074828 (Reference) | Part A: 250 mg LY3074828 (Test 1)
Number analyzed (Participants) | 18 | 18
units on a scale | 4.16 [2.88 to 6.01] | 3.04 [2.10 to 4.39]
Statistical Analysis 1: Comparison: Part A: 250 mg LY3074828 (Reference) vs Part A: 250 mg LY3074828 (Test 1); Test type: Superiority; Ratio of Geometric Least Squares Means = 0.73, 90% CI 2-sided [0.43 to 1.23]

5. Primary Outcome: Part B: Short Form McGill Pain Questionnaire (SF-MPQ) Total Score (Including VAS Score) For 250 mg LY3074828 Slow Versus Fast
Description: Pain was assessed by the SF-MPQ and quantified using the validated VAS where 0mm represented "no pain" and 100mm represented "worst possible pain". The SF-MPQ total score ranges from 0 to 45 (the higher the total score, the more pain experienced). LS mean was calculated using linear fixed-effects model with treatment (Test 2 or Test 3) as a fixed effect. Model: Log (Score+1) = Treatment + Random Error.
Time Frame: Day 1, 0 hour
Population: All participants who received a dose of LY3074828 whether or not they completed all protocol requirements.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: units on a scale
Groups:
- Part B: 250 mg LY3074828 (Test 2): Test 2: 250 mg LY3074828 administered subcutaneous (SC) as solution formulation in an auto-injector at slow speed targeting an approximately 13-second injection time on day 1.
- Part B: 250 mg LY3074828 (Test 3): Test 3: 250 mg LY3074828 administered subcutaneous (SC) as solution formulation in an auto-injector at fast speed targeting an approximately 5-second injection time on day 2.
Arm/Group | Part B: 250 mg LY3074828 (Test 2) | Part B: 250 mg LY3074828 (Test 3)
Number analyzed (Participants) | 9 | 9
units on a scale | 5.06 [3.48 to 7.36] | 4.96 [3.41 to 7.22]
Statistical Analysis 1: Comparison: Part B: 250 mg LY3074828 (Test 2) vs Part B: 250 mg LY3074828 (Test 3); Test type: Other; Ratio of geometric least squares mean = 0.98, 90% CI 2-sided [0.58 to 1.67]

6. Primary Outcome: Part B: Short Form McGill Pain Questionnaire (SF-MPQ) Total Score (Including VAS Score) For 125 mg LY3074828 Slow Versus Fast
Description: Pain was assessed by the SF-MPQ and quantified using the validated VAS where 0mm represented "no pain" and 100mm represented "worst possible pain". The SF-MPQ total score ranges from 0 to 45 (the higher the total score, the more pain experienced). LS mean was calculated using linear fixed-effects model with treatment (Test 4 or Test 5) as a fixed effect. Model: Log (Score+1) = Treatment + Random Error.
Time Frame: Day 1, 0 hour
Population: All participants who received a dose of LY3074828 whether or not they completed all protocol requirements.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: units on a scale
Groups:
- Part B: 125 mg LY3074828 (Test 4): Test 4: 125 mg LY3074828 administered SC as solution formulation in an auto-injector at slow speed targeting an approximately 7-second injection time on day 1.
- Part B: 125 mg LY3074828 (Test 5): Test 5: 125 mg LY3074828 administered SC as solution formulation in an auto-injector at fast speed targeting an approximately 4.5-second injection time on day 2
Arm/Group | Part B: 125 mg LY3074828 (Test 4) | Part B: 125 mg LY3074828 (Test 5)
Number analyzed (Participants) | 9 | 9
units on a scale | 4.36 [3.00 to 6.35] | 3.07 [2.11 to 4.47]
Statistical Analysis 1: Comparison: Part B: 125 mg LY3074828 (Test 4) vs Part B: 125 mg LY3074828 (Test 5); Test type: Other; Ratio of geometric least squares mean = 0.70, 90% CI 2-sided [0.41 to 1.20]

ADVERSE EVENTS:
Time Frame: Baseline Up To Day 88
Description: All participants who received at least one dose of study drug.
Arm/Group | Part A: 250 mg LY3074828 (Reference) | Part A: 250 mg LY3074828 (Test 1) | Part B: 250 mg LY3074828 (Test 2) | Part B: 250 mg LY3074828 (Test 3) | Part B: 125 mg LY3074828 (Test 4) | Part B: 125 mg LY3074828 (Test 5)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 6/18 | 1/18 | 5/18 | 1/18 | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 250 mg LY3074828 (Reference) (N=18) | Part A: 250 mg LY3074828 (Test 1) (N=18) | Part B: 250 mg LY3074828 (Test 2) (N=18) | Part B: 250 mg LY3074828 (Test 3) (N=18) | Part B: 125 mg LY3074828 (Test 4) (N=18) | Part B: 125 mg LY3074828 (Test 5) (N=18)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT03456713/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT03456713/SAP_001.pdf